CLINICAL TRIAL: NCT05254392
Title: The Impact of Pharmacists' Interventions on Blood Pressure Among Patients With Chronic Kidney Disease: a Randomized Controlled Trial
Brief Title: Pharmacists' Interventions to Improve Blood Pressure in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maiduguri (Other)
Responsible Party: Principal Investigator, Roland Nnaemeka Okoro, Principal Investigator, University of Maiduguri
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PharmBP
Record Dates: First submitted 2022-02-05; First posted 2022-02-24 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Chronic Kidney Diseases
Keywords: Blood pressure; Chronic Kidney Disease; Home blood pressure self-monitoring; Nigeria; Pre-dialysis; Pharmacists' interventions
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were blinded to the profession of the investigators and study arms, while outcome assessors were blinded to the interventions and study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants in the UC arm received the usual/conventional care offered by the hospitals which included: hospital visits on appointment or a sick day, consultations with the physicians, prescription of drugs and routine laboratory tests, review of diagnosis and medications, refilling of prescriptions by patients and referral.
- Pharmacists' Intervention (Experimental): Participants in the PI arm received routine usual care plus pharmacists' interventions for 12 months. The PI arm received usual care plus face-to-face education on CKD, hypertension as a co-morbidity and its management, and antihypertensive medication adherence at baseline (group education), 6 months and 12 months (individualized according to each patient's needs), CKD patient educational infographic leaflet at baseline, a calibrated sphygmomanometer digital BP monitor (Chidalex®) for HSMBM, a BP logbook at baseline for the recording of BP values daily and hands-on training on BP self-measurement. Also, antihypertensive medication adherence and HSMBM reminder cell phone text messages were sent biweekly throughout the trial period, while phone-in inquiries from the participants and phone-out reinforcement interventions were utilized throughout the trial period
  Interventions: Device: Digital BP monitor (Chidalex®)

INTERVENTIONS:
Device: Digital BP monitor (Chidalex®) — Interventions were provided in groups of 4 - 10 participants after data collection at baseline while reinforcing individualized interventions were provided during subsequent visits to the research clinic for follow-up at 6 months and 12 months. Medication reminder text messages were delivered to each participant biweekly.
  Other Names: Chronic Kidney Education; Medication adherence reminder text messages; Other tele-interventions
  Arms: Pharmacists' Intervention

SUMMARY:
The aims of the study were to determine whether pharmacists' interventions combining patient home-based self-measured BP monitoring improve blood pressure reduction and control compared with usual care in chronic kidney disease (CKD) patients

DETAILED DESCRIPTION:
This is a prospective randomized two-group pharmacist-led interventional study that was conducted in two public nephrology clinics. The study involved the introduction of pharmaceutical care to improve blood pressure and adherence to the prescribed medications among patients with chronic kidney disease (CKD).

Recruited patients were randomly divided into two groups; the intervention group and the control group, with baseline evaluation of outcomes measured.

The Control group was provided with usual care. An intervention group was provided in addition to the usual care, face-to-face education on CKD, hypertension as a co-morbidity and its management, and antihypertensive medication adherence at baseline (group education), 6 months and 12 months (individualized according to each patient's needs), CKD patient educational infographic leaflet at baseline, a calibrated sphygmomanometer digital blood pressure monitor (Chidalex®) for home-based self-measured BP monitoring, a BP logbook at baseline for the recording of blood pressure values daily and hands-on training on BP self-measurement. Also, antihypertensive medication adherence and home-based self-measured BP monitoring, reminder cell phone text messages were sent biweekly throughout the trial period, while phone-in inquiries from the participants and phone-out reinforcement interventions were utilized throughout the trial period.

Both groups were followed for a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* CKD stages 1 - 4,
* Voluntary written informed consent,
* Willingness to abide by the rules of trial, and
* Availability during the trial duration

Exclusion Criteria:

* Patients with acute renal failure,
* CKD stage 5,
* Pregnant or lactating women,
* Post-renal transplant patients,
* Patients with HIV infection,
* Critically ill patients or patients known to have cognitive impairment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in mean blood pressure | 6 months and 12 months
  Changes in both mean systolic and diastolic blood pressure.overtime were determined
Changes in blood pressure control | 6 months and 12 months
  Changes in the proportion of participants with both controlled systolic and diastolic blood pressure less than 130/80 mmHg overtime were measured

SECONDARY OUTCOMES:
Changes in mean antihypertensive medication adherence | 6 months and 12 months
  Antihypertensive medication adherence was determined using the 4-item Morisky-Green-Levine (MGL) scale. The response was scored as follows: a "yes" response was scored one point and zero to a "no" response. The total score ranged from zero to four. Adherence levels were then categorized into three based on the total score. Zero, 1 - 2, and 3 - 4 were classified as high adherence, moderate adherence, and low adherence, respectively. Lower scores mean a better outcome.
Changes in mean serum creatinine levels | 6 months and 12 months
  Participants' blood samples were analyzed for creatinine levels
Participants' satisfaction with care received | 12 months
  The Patient Satisfaction with Pharmacist Services Questionnaire (PSPSQ) 2.0 (Sakharkar et al., 2015) was used to assess patient satisfaction with care received. The participants' responses to items 1-19 were scored 4 points, 3 points, 2 points, and 1 point, respectively for "strongly agreed", "agree", "disagree", and "strongly disagree". However, item 20 was also scored 4 points, 3 points, 2 points, and 1 point, respectively for "exceeded your expectation", "met your expectation", "did not meet your expectation", and "I had no expectation". For the quality of care domain, minimum value is 1 and maximum value is 40, For interpersonal relationship domain, minimum value is 1 and maximum value is 24. For overall satisfaction domain, minimum value is 1 and maximum value is 16.Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Roland N Okoro, PhD, Principal Investigator — University of Maiduguri
Locations (2):
- Nigeria (2):
  - State Specialist Hospital, Maiduguri, Borno State
  - University of Maiduguri Teaching Hospital, Maiduguri, Borno State

IPD SHARING:
Plan to Share IPD: No